CLINICAL TRIAL: NCT05706688
Title: Effect of Regional Versus General Anesthesia on Thirty-day Outcomes Following Carotid Endarterectomy: a Matched-pairs Cohort Study.
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Zhiyi Zuo, MD, Principal Investigator, University of Virginia
Other Study IDs: HSRZOKZZ
Record Dates: First submitted 2023-01-21; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Regional Anesthesia Morbidity; Carotid Artery Diseases; Perioperative/Postoperative Complications
MeSH Terms: conditions — Carotid Artery Diseases; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regional anesthesia: 4,152 patients undergoing elective carotid endarterectomy under regional anesthesia
  Interventions: Procedure: Anesthetic technique (regional versus general)
- General anesthesia: 4,152 matched controls undergoing elective carotid endarterectomy under general anesthesia
  Interventions: Procedure: Anesthetic technique (regional versus general)

INTERVENTIONS:
Procedure: Anesthetic technique (regional versus general) — Anesthetic technique (regional versus general)

SUMMARY:
The goal of this observational study is to assess the effect of regional versus general anesthesia on carotid endarterectomy thirty-day outcomes. The main questions it aims to answer are:

* Is regional anesthesia associated with lower incidence of major morbidity and mortality?
* Is regional anesthesia associated with lower incidences of secondary adverse events?

Participants will be sampled from the 2015-2019 American College of Surgeons National Surgical Quality Improvement Program

ELIGIBILITY:
Inclusion Criteria:

* Elective, non-emergent cases
* Regional anesthesia
* General anesthesia

Exclusion Criteria:

* Concurrency in procedures
* Acute kidney injury (preoperative)
* End-stage renal disease (preoperative)
* Metastatic disease (preoperative)
* Wound infection (preoperative)
* Sepsis (preoperative)
* ASA 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elective carotid endarterectomy patients, ACS-NSQIP 2015-2019
Sampling Method: Non-Probability Sample
Enrollment: 37204 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Major morbidity and mortality | Thirty days
  Stoke, myocardial infarction, or death

SECONDARY OUTCOMES:
Minor morbidity | Thirty days
  Reintubation, prolonged (>48 hour) ventilator dependence, pneumonia, deep venous thrombosis, pulmonary embolism, superficial surgical site infection (SSI), deep incisional SSI, organ space SSI, wound dehiscence, sepsis, septic shock, acute kidney injury, and progressive renal insufficiency
Bleeding events | Thirty days
  Requiring transfusion
Unplanned resource utilization | Thirty days
  Unplanned readmission and unplanned reoperation
Mortality | Thirty days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyi Zuo, MD, PhD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: Yes
American College of Surgeons National Surgical Quality Improvement Program and the hospitals participating in the ACS NSQIP are the source of the data used herein. The Participant Use Data File (PUF) is a Health Insurance Portability and Accountability Act (HIPAA)-compliant data file containing cases submitted to the American College of Surgeons National Surgical Quality Improvement Program®. To request a copy of the PUF, individuals (data recipients) must agree to comply with the terms and conditions set forth in the Data Use Agreement, provide contact information, and complete a short online questionnaire. Once the information provided by the data recipient is received and processed by ACS NSQIP staff, a website address will be submitted electronically to the data recipient. The data recipient will then have 10 days (240 hours) to visit the website and download the data file.

REFERENCES:
- [Derived] Kline LA, Kothandaraman V, Knio ZO, Zuo Z. Effect of regional versus general anesthesia on thirty-day outcomes following carotid endarterectomy: a cohort study. Int J Surg. 2023 May 1;109(5):1291-1298. doi: 10.1097/JS9.0000000000000356. PMID 37057905
- Available data/document: Individual Participant Data Set — https://www.facs.org/quality-programs/data-and-registries/acs-nsqip/participant-use-data-file/ — American College of Surgeons National Surgical Quality Improvement Program and the hospitals participating in the ACS NSQIP are the source of the data used herein. The Participant Use Data File (PUF) is a Health Insurance Portability and Accountability Act (HIPAA)-compliant data file containing cases submitted to the American College of Surgeons National Surgical Quality Improvement Program®. To request a copy of the PUF, individuals (data recipients) must agree to comply with the terms and conditions set forth in the Data Use Agreement, provide contact information, and complete a short online questionnaire. Once the information provided by the data recipient is received and processed by ACS NSQIP staff, a website address will be submitted electronically to the data recipient. The data recipient will then have 10 days (240 hours) to visit the website and download the data file.